CLINICAL TRIAL: NCT04697342
Title: Nantou Hospital, Ministry of Health and Welfare, Taiwan
Brief Title: Nantou Hospital, Regional Teaching Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wen-Yi Chao (Other Government)
Responsible Party: Sponsor-Investigator, Wen-Yi Chao, Principal Investigator, Nantou Hospital
Organization: Nantou Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NantouH
Record Dates: First submitted 2020-12-29; First posted 2021-01-06 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Knowledge, Attitudes, Practice; Self Efficacy; Learning
Keywords: continued learning; Knowledge, Attitudes, Practice; self efficacy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: The head nurse is blinded, and the unit nurses are randomly arranged according to the unit to participate in any education training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIS with pressure injury(PI) education (Active Comparator): Clinical nurses use Nursing information system(NIS) to log in nursing records every day, and pressure injury (PI) education pops out of the NIS window for teaching
  Interventions: Behavioral: strategy of education
- NIS with PI education, and microvideo (Active Comparator): In addition to the built-in PI education in the NIS that nurses use every day, it also provides a flipped digital learning plan course unit, which can be self-study courses anytime, anywhere, without being restricted by time and space. And hold a 4-hour physical course for participants.
  Interventions: Behavioral: strategy of education
- NIS with PI education, and workshop (Experimental): In addition to the built-in PI education in the NIS that nurses use every day, an 8-hour physical course is also provided.
  Interventions: Behavioral: strategy of education

INTERVENTIONS:
Behavioral: strategy of education — one of the strategies is microvideo with nursing information system(NIS); another of the strategies is workshop with NIS.
  NIS of PI education is the routine education

SUMMARY:
The incidence of crush is one of the important indicators of the quality of health care in various medical institutions in the world. The Taiwan Hospital Evaluation and Medical Quality Council (referred to as the Medical Policy Council) listed crush as a quality indicator of clinical care in 2011 (Taiwan Clinical Effectiveness indicator system, 2011), the incidence of crush is also a sensitive indicator of nursing care.

The purpose of this study: based on the nursing of crushed wounds, intervene in education and training courses, and add elements of flipped learning, to evaluate the effectiveness of KAP (knowledge, attitude, practice) and self efficacy of nursing staff for learning crushed nursing.

DETAILED DESCRIPTION:
The incidence of crush is one of the important indicators of the quality of health care in various medical institutions in the world. The Taiwan Hospital Evaluation and Medical Quality Council (referred to as the Medical Policy Council) listed crush as a quality indicator of clinical care in 2011 (Taiwan Clinical Effectiveness indicator system, 2011), the incidence of crush is also a sensitive indicator of nursing care, reflecting the effectiveness of the structure, process and results of nursing care (Cai, Zheng, Liu, 2011). Reducing the incidence of crush has been the goal of the joint efforts of health care institutions. In 2008, the US CMS announced that it would stop paying for the treatment of crushed patients in hospitals, allowing medical institutions to pay more attention to the prevention of crushing, so many promote the quality of medical care The organizations have put forward relevant strategies, including the announcement of evidence-based tools for predicting and evaluating crush injuries, guidelines on the classification and prevention of crush injuries, and training materials for crush education (Agency for Healthcare Research and Quality, 2014; Edsberg et al ., 2016; Institute for Healthcare Improvement, 2017). The occurrence of pressure injury can be prevented. Many studies have explored the reasons why nursing staff cannot implement the behaviors of pressure injury prevention. The results show that the common obstacles are the lack of time and manpower of nursing staff, lack of relevant education and training, and failure to provide standard operations. Routine, physicians did not participate, etc. (Jankowski & Nadzam, 2011; Moore & Price, 2004; Worsley, Clarkson, Bader, & Schoonhoven, 2016).

At the same time, many researchers have explored the impact of various education and training methods on nursing staff's cognition, behavior and attitude related to the prevention and treatment of crush. They can all prove that education and training measures can significantly improve nursing staff's cognition. These important changes must be carefully considered as to what learning or training methods should be used to provide first-line nursing staff to familiarize them with and correctly perform practical operations. Clinical nurses are faced with ever-changing patient situations. The goal of learning is not only to transfer knowledge to enhance cognition, but more importantly, how to transform knowledge into clinical practice skills and provide clinical decision-making with appropriate care measures in response to different situations. Ability, teaching must use multiple strategies to achieve this goal, providing a real and interactive learning environment, allowing nurses to participate in operational activities in a simulated real environment, repeatedly learning related knowledge and techniques, and strengthen the proficiency of clinical applications And to build consensus on care can improve the quality of work (Norman, 2012).

The purpose of this study: based on the nursing of crushed wounds, intervene in education and training courses, and add elements of flipped learning, to evaluate the effectiveness of KAP (knowledge, attitude, practice) and self efficacy of nursing staff for learning crushed nursing.

ELIGIBILITY:
Inclusion Criteria:

* Have a nurse practitioner license in Nantou Hospital
* work as a clinician

Exclusion Criteria:

* Nursing student

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge of pressure ulcer | 2days
  The section measure nurses" knowledge regarding pressure ulcer prevention, staging, and wound description. The researcher used a known, public and validated available tool of Pieper Pressure Ulcer Knowledge Test. (Pieper and oton,1959). The tool has 39 items of yes, no, I don"t know.
  =90%-100% showed a very high level of knowledge, 80%-89,99% showed a high level of knowledge, 70%-79, 99% showed a moderate level of knowledge, 60%-69, 99% showed a low level of knowledge, And a percentage below 60% showed a very low level of knowledge.
Attitude of pressure ulcer | 2days
  The section has 11 items describing the nurses "attitudes regarding pressure ulcer prevention. The researcher used the validate "Staff Attitude Scale" adapted from a scale used by Moore and Price which is also an a scale open to the public (to use the instrument does not require permission). Each item has 5 point scoring system ranging from strongly agree to strongly disagree." Here, "strongly disagree" = 5 points, "disagree" = 4 points, "Neither agree nor disagree"=3 points, Agree=2 points and "Strongly agree"=1 point. (Moore Z, Price P, 2004).
Practice of pressure ulcer | 2days
  This tool originally consisted of multiple-choice questions with "Yes", "no", "responsible person" and "comment" as options but after adaptation, only "yes" or "no" remained as options.
  The McDonald"s standard of learning outcome was used to interpret the level of practice as either low or high as follow.(McDonald, 2002): A percentage of 60% indicated a very low level of practices, A percentage of 60%-69,99% indicated a low level of practices , A percentage of 70%-79,99% indicated a moderate level of practices, A percentage of 80%-89, 99% indicated a high level of practices, A percentage of 90%-100% indicated a very high-level of practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantou Hospital, Nantou City, Taiwan

IPD SHARING:
Plan to Share IPD: No